CLINICAL TRIAL: NCT01476722
Title: Lens Wearing Experience and Biocompatibility With OPTI-FREE® PureMoist® Multi-Purpose Disinfecting Solution (OFP MPDS) in Silicone Hydrogel and Soft Contact Lens Wearers (US)
Brief Title: Lens Wearing Experience and Biocompatibility of a Multi-Purpose Disinfecting Solution (MPDS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: RDG-11-149
Record Dates: First submitted 2011-11-18; First posted 2011-11-22 (Estimated); Results first posted 2012-11-19 (Estimated); Last update posted 2012-11-19 (Estimated); Status verified 2012-11

CONDITIONS: Healthy
Keywords: Silicone Hydrogel; Soft Contact Lenses; Multi-Purpose Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- OPTI-FREE PureMoist (Experimental): OPTI-FREE PureMoist multipurpose disinfecting solution used with study contact lenses on a daily wear basis for 30 days
  Interventions: Device: OPTI-FREE PureMoist multipurpose disinfecting solution

INTERVENTIONS:
Device: OPTI-FREE PureMoist multipurpose disinfecting solution — FDA-approved, multipurpose disinfecting solution used as indicated for cleaning, rinsing, reconditioning, disinfecting, and storing silicone hydrogel and soft contact lenses on a daily wear basis for 30 days

SUMMARY:
The purpose of this study was to evaluate the efficacy of a new multipurpose disinfecting solution in silicone hydrogel and soft contact lens wearers.

ELIGIBILITY:
Inclusion Criteria:

* Wear silicone hydrogel or traditional soft contact lenses on a daily wear basis, (a minimum of 8 hours per day) for at least one month prior to Visit 1;
* Habitual use of a multi-purpose solution containing PHMB for at least 30 days prior to Visit 1;
* Vision correctable to 20/30 (Snellen) or better in each eye at distance with pre-study lenses at Visit 1;
* Read, sign, and date IRB-approved informed consent and privacy document;
* Be generally healthy and have normal ocular health;
* Willing to follow the study procedures and visit schedule;
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria

* Wear lenses on an extended wear basis during the study;
* Known sensitivity or intolerance to PHMB, POLYQUAD, or ALDOX preserved lens care products;
* Monocular subject;
* Requirestoric or multifocal contact lenses;
* Use of additional lens care products other than a PHMB multi-purpose solution such as daily or enzyme cleaners within the one week prior to Visit 1;
* Use of topical ocular over-the-counter (OTC) or prescribed topical ocular medications, with the exception of rewetting drops, within 7 days prior to Visit 1;
* Any abnormal ocular condition observed during the Visit 1 Slit-lamp examination;
* Ocular surgery within the 12 months prior to Visit 1;
* Use of any systemic medication which has known or expected ocular or systemic side effects at Visit 1, that in the clinical judgment of the investigator, could affect the subject's participation in this study;
* Any systemic disease at Visit 1 that may affect the eye or be exacerabated by use of contact lenses or contact lens solutions or which could prevent subjects from wearing their lenses at least 8 hours per day;
* Participation in any clinical study within 30 days of Visit 1;
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2011-06; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Contact Alcon Call Center for Trial Locations, Fort Worth, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 5 US study centers.
Period: Overall Study
Arm/Group | OPTI-FREE PureMoist
Started | 125
Completed | 124
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | OPTI-FREE PureMoist
Number analyzed (Participants) | 124
Age Continuous [Mean (Standard Deviation); unit: years] — Baseline characteristics are presented for all enrolled subjects who received test article and had at least 1 on-therapy visit (ITT): 124.
  years | 32.2 (11.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89
  Male | 35
Region of Enrollment [Number; unit: participants]
  United States | 124

OUTCOME MEASURES:

1. Primary Outcome: Corneal Fluorescein Staining Type at Baseline
Description: Corneal staining type was assessed by the investigator for each of 5 regions of the cornea, i.e., four quadrants plus central. The investigator instilled fluorescein dye and examined the cornea with a slit lamp, i.e., biomicroscope and a yellow filter. Corneal staining type was recorded on a 5-point scale for each region: 0-none; 1-micropunctate; 2-macropunctate; 3-coalesced macropunctate; 4-patch (>/= 1mm). The five regions were summed, for a maximum score of 20. A lower score represents a more desirable outcome.
Time Frame: Day 0 (Baseline)
Population: Intent-to-treat. All enrolled subjects who received test article and had at least 1 on-therapy visit.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OPTI-FREE PureMoist
Number analyzed (Participants) | 124
Units on a scale | 1.7 (1.38)

2. Primary Outcome: Corneal Fluorescein Staining Type at Day 30
Description: as for outcome 1
Time Frame: Day 30
Population: Intent-to-treat. All enrolled subjects who received test article and had at least 1 on-therapy visit.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OPTI-FREE PureMoist
Number analyzed (Participants) | 124
Units on a scale | 0.7 (0.94)

3. Primary Outcome: Corneal Fluorescein Staining Area at Baseline
Description: Corneal staining was assessed by the investigator for each of five regions of the cornea, i.e., four quadrants plus central. The investigator instilled fluorescein dye and examined the cornea with a slit lamp, i.e., biomicroscope and a yellow filter. The area (extent) of corneal staining for each of the five areas was estimated [i.e., 0% (no staining in the region) to 100% (staining covers entire region)], for a maximum score of 100% per eye. A lower score represents a more desirable outcome.
Time Frame: Day 0 (Baseline)
Population: Intent-to-treat. All enrolled subjects who received test article and had at least 1 on-therapy visit.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OPTI-FREE PureMoist
Number analyzed (Participants) | 124
Units on a scale | 5.6 (9.34)

4. Primary Outcome: Corneal Fluorescein Staining Area at Day 30
Description: as for outcome 3
Time Frame: Day 30
Population: Intent-to-treat. All enrolled subjects who received test article and had at least 1 on-therapy visit.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OPTI-FREE PureMoist
Number analyzed (Participants) | 124
Units on a scale | 1.4 (2.41)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study (e.g., 4 months).
Description: The safety population includes all enrolled and exposed subjects. Both volunteered and elicited adverse events were collected, monitored, and evaluated through the study.
Arm/Group | OPTI-FREE PureMoist
Serious Adverse Events (participants affected / at risk) | 0/125
Other Adverse Events (participants affected / at risk) | 0/125

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.